CLINICAL TRIAL: NCT00895037
Title: Pharmacovigilance Evaluation Of Refacto Af (Registered) In Germany And Austria
Brief Title: Study Evaluating Pharmacovigilance Of Refacto AF
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3082B2-4420; B1831016 (Other: Alias Study Number)
Record Dates: First submitted 2009-05-01; First posted 2009-05-07 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2017-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; recombinant factor VIII SQ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients treated with Refacto AF
  Interventions: Drug: ReFacto AF (Moroctocog alfa)

INTERVENTIONS:
Drug: ReFacto AF (Moroctocog alfa) — Patients will be treated with intravenous infusion of ReFacto AF per dosing and frequency as prescribed by the subjects' treating physician. ReFacto AF® will be prescribed in the context of routine clinical practice in Germany and Austria, respectively

SUMMARY:
The purpose of this observational study is to describe the incidence of adverse events among patients treated with Refacto AF in usual health care settings in Germany and Austria.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A of any severity already receiving or starting treatment with ReFacto AF.

Exclusion Criteria:

* Patients with Hemophilia A treated with a product other than Refacto AF.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2009-07-17 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Austria (3):
  - LKH - Univ. Klinikum Graz,Abt. fur Hamatologie, Graz
  - Allgemeines Krankenhaus Linz, Kinderklinik, Linz
  - Universitaetsklinik fuer Innere Medizin 1, Vienna
- Germany (21):
  - Sonnengesundheitszentrum, München, Bavaria
  - Werlhof-Institut für Haemostaseologie GmbH, Hanover, Lower Saxony
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum Bremen Mitte, Bremen
  - CRC Coagulation Research Centre GmbH, Duisburg
  - Universitaetsklinikum Duesseldorf, Klinik f. Kinder-Onkologie, Haematologie u. Klinische Immunologie, Düsseldorf
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Praxis zur Diagnostik und Therapie Von Blutgerinnungstoerungen, Frankfurt A. M.
  - Praxis fur Kinder- und Jugendmedizin, Grünwald
  - Medizinische Hochschule Hannover, Hanover
  - SRH Kurpfalzkrankenhaus Heidelberg, Heidelberg
  - Donaustrasse 78, Memmingen
  - Praxis Dr. Autenrieth, Metzingen
  - Hämophilie-Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Stauferklinikum Schwaebisch Gmuend, Mutlangen
  - Institut for Thrombophilia and Hemastaseologie, Münster
  - Universität Regensburg, Regensburg
  - Asklepios Fachklinikum Stadtroda GmbH, Stadtroda
  - Klinikum Stuttgart, Stuttgart
  - Universitaetsklinik fuer Kinder- und Jugendmedizin, Tübingen
  - Stiftung Deutsche Klinik fur Diagnostik GmbH, Wiesbaden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-4420&StudyName=Study%20Evaluating%20Pharmacovigilance%20Of%20Refacto%20AF

RESULTS

PARTICIPANT FLOW:
Groups:
- ReFacto AF: On Demand Treatment: Participants were treated with intravenous (IV) injection of ReFacto AF whenever they had a bleeding episode, as a part of routine clinical practice at a dose and frequency prescribed by treating physician (with a mean recommended dose of 23.0 ± 8.0 international units per kilogram [IU/kg]). Participants were observed for up to a maximum duration of 87 months in this study.
- ReFacto AF: Prophylaxis Treatment: Participants were treated prophylactically with a regular IV injection of ReFacto AF to prevent any bleeding episode at a dose and frequency prescribed by treating physician (with a mean recommended dose of 26.7 ± 8.4 IU/kg). Participants were observed for up to a maximum duration of 87 months in this study.
- ReFacto AF: Intermediate Prophylaxis Treatment: Participants had intermediate prophylaxis (regular dosing with drug at a low dose than the defined prophylactic treatment) treatment with a regular IV injection of ReFacto AF to prevent any bleeding episode at a dose and frequency prescribed by treating physician (with a mean recommended dose of less than [>] 26.7 ± 8.4 IU/kg). Participants were observed for up to a maximum duration of 87 months in this study.
Period: Overall Study
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Started | 22 | 77 | 2
Completed | 22 | 75 | 1
Not Completed | 0 | 2 | 1
Not completed — Death | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of ReFacto AF.
Groups:
- Total: Total of all reporting groups
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment | Total
Number analyzed (Participants) | 22 | 77 | 2 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (20.2) | 18.5 (12.4) | 62.0 (7.1) | 22.7 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 22 | 77 | 2 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; cancer; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to last visit (up to 87 months) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline until last visit (up to 87 months)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of ReFacto AF.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 22 | 77 | 2
participants
  AEs | 15 | 59 | 2
  SAEs | 7 | 25 | 2

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; cancer; congenital anomaly. AEs included both serious and non-serious adverse events. Relatedness of AEs with Refacto AF was assessed by the investigator.
Time Frame: Baseline until last visit (up to 87 months)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of ReFacto AF.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 22 | 77 | 2
participants
  AEs | 2 | 7 | 0
  SAEs | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Factor VIII (FVIII) Inhibitor Development as Measured by the Nijmegen-Modified Bethesda Assay
Description: FVIII inhibitor development was defined as measured inhibitor titer of greater than (>) 0.6 Bethesda Units (BU) using the Nijmegen-modified Bethesda assay.
Time Frame: Baseline until last visit (up to 87 months)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of ReFacto AF.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 22 | 77 | 2
participants | 1 | 2 | 0

4. Primary Outcome: Mean Total Number of Bleeding Episodes in Participants
Description: Participants documented all bleeding episodes in a diary during the study.
Time Frame: Baseline until last visit (up to 87 months)
Population: Effectiveness analysis set =participants registered in study and had at least 1 dose of ReFacto AF documented by participants diary entries. Participant's registration included confirmation of obtained participant's informed consent from the physician. Here, 'N' (number of participants analyzed) = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: bleeding episodes
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 17 | 74 | 2
bleeding episodes | 71.2 (73.3) | 15.4 (14.7) | 68.5 (31.8)

5. Secondary Outcome: Mean Total Number of Bleeding Episodes Per Year in Participants
Description: Participants documented all bleeding episodes in a diary during the study. Mean total number of bleeding episodes per year was calculated as: mean total number of bleeding episodes divided by duration of observation period (in years) for bleeding documentation.
Time Frame: Baseline until last visit (up to 87 months)
Population: Effectiveness analysis set =participants registered in study and had at least 1 dose of ReFacto AF documented by participants diary entries. Participant's registration included confirmation of obtained participant's informed consent from the physician. Here, 'N' =participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: bleeding episodes per year
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 17 | 74 | 2
bleeding episodes per year | 18.6 (19.6) | 5.1 (5.8) | 13.4 (0.5)

6. Secondary Outcome: Number of Participants With Change From Baseline Status in Days Missed From School or Work
Description: Change from baseline status in days missed from school or work was categorized in 3 categories: Improvement, unchanged and worsening. Improvement defined as a decrease in number of days missed by participants from school/work as compared to baseline; worsening was defined as an increase in number of days missed by participants from school/work as compared to baseline; unchanged was defined as no change in number of days missed by participants from school/work as compared to baseline. In this outcome measure, number of participants with change from baseline status (as improved, worsen, unchanged) in days missed from school/work were reported.
Time Frame: Baseline until last visit (up to 87 months)
Population: Analysis was performed on effectiveness analysis set. Here, 'N' signifies those participants who were evaluable for this outcome measure. For this outcome measure, data for Refacto AF: intermediate prophylaxis treatment arm could not be analyzed since all participants of this arm were neither working nor school going.
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment
Number analyzed (Participants) | 11 | 60
participants
  Improvement | 4 | 25
  Unchanged | 4 | 29
  Worsening | 3 | 6

7. Secondary Outcome: Participant Assessment of Satisfaction With Treatment Handling
Description: Participants evaluated their satisfaction with handing (administration) of Refacto AF and rated it in 4 categories as: very satisfied, satisfied, unsatisfied and very unsatisfied.
Time Frame: End of study visit (any time up to 87 months)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 18 | 74 | 2
participants
  Very satisfied | 13 | 42 | 0
  Satisfied | 5 | 28 | 2
  Unsatisfied | 0 | 4 | 0
  Very unsatisfied | 0 | 0 | 0

8. Secondary Outcome: Investigator Assessment of Treatment Satisfaction of Participants
Description: Investigator assessed the treatment satisfaction of participants and categorized as very satisfied, satisfied, unsatisfied, or very unsatisfied.
Time Frame: End of study visit (any time up to 87 months)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Number analyzed (Participants) | 17 | 74 | 2
participants
  Very satisfied | 13 | 44 | 0
  Satisfied | 4 | 29 | 2
  Unsatisfied | 0 | 1 | 0
  Very unsatisfied | 0 | 0 | 0

ADVERSE EVENTS:
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | ReFacto AF: On Demand Treatment | ReFacto AF: Prophylaxis Treatment | ReFacto AF: Intermediate Prophylaxis Treatment
Serious Adverse Events (participants affected / at risk) | 7/22 | 25/77 | 2/2
Other Adverse Events (participants affected / at risk) | 14/22 | 56/77 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto AF: On Demand Treatment (N=22) | ReFacto AF: Prophylaxis Treatment (N=77) | ReFacto AF: Intermediate Prophylaxis Treatment (N=2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Oesophageal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Inhibiting antibodies positive (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint adhesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0
Antisocial personality disorder (Psychiatric disorders) | 1 | 0 | 0
Apathy (Psychiatric disorders) | 1 | 0 | 0
Personality disorder (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReFacto AF: On Demand Treatment (N=22) | ReFacto AF: Prophylaxis Treatment (N=77) | ReFacto AF: Intermediate Prophylaxis Treatment (N=2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Platelet disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Factor V deficiency (Congenital, familial and genetic disorders) | 0 | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Catheter site phlebitis (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Febrile infection (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Herpes dermatitis (Infections and infestations) | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0
Scarlet fever (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 11 | 0
Exposure via father (Injury, poisoning and procedural complications) | 1 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 17 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Genital injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 4 | 14 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 8 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 7 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 13 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 1 | 3 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 4 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 4 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 3 | 16 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 4 | 0
Colonoscopy (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 12 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 15 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dental care (Surgical and medical procedures) | 1 | 1 | 0
Ear operation (Surgical and medical procedures) | 0 | 1 | 0
Eye operation (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 3 | 0
Wedge resection toenail (Surgical and medical procedures) | 0 | 0 | 1
Wisdom teeth removal (Surgical and medical procedures) | 1 | 3 | 0
Haematoma (Vascular disorders) | 2 | 5 | 0
Haemorrhage (Vascular disorders) | 1 | 6 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures as primary and secondary was based on the study team's discretion, as it was not specified in source documents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.